CLINICAL TRIAL: NCT01578941
Title: An Investigation of the Safety and Utility of Treximet in the Treatment of Menstrual Migraine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Principal Investigator, J. Ivan Lopez, MD, Professor of Neurology, University of Alabama at Birmingham
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: Treximet-UAB-Glaxo
Record Dates: First submitted 2012-01-05; First posted 2012-04-17 (Estimated); Last update posted 2012-11-01 (Estimated); Status verified 2012-10

CONDITIONS: Menstrual Migraine
Keywords: menstrual migraine; migraine; treximet
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Other: Diary
- Treximet (Active Comparator)
  Interventions: Other: Diary

INTERVENTIONS:
Other: Diary — Each subject will be asked to keep a careful headache diary (appendix B) , and in that diary she will record onset and cessation of menstrual flow, days of menstrual headache (and "migraine" headache, specifically) experienced, days of functionally incapacitating headache experienced, any abortive/symptomatic medications taken, any days of work-related absenteeism (>4 hrs) related to acute MM headache and any unscheduled visits to a medical facility for acute treatment of MM.

SUMMARY:
The study is to primarily investigate whether Treximet® (Imitrex RT/naproxen sodium 500mg) taken at the first onset of menstrual migraine will both terminate the acute headache and assist in preventing headache recurrence and the need for repeat abortive therapy over the ensuing days of menses.

ELIGIBILITY:
Inclusion Criteria:

1. Actively and regularly cycling females age 19 years or greater.
2. Normal (for subject) menses within 6 weeks prior to randomization
3. History of migraine of ≤ 1 years duration by International Classification of Headache Disorders (ICHD) criteria
4. History of menstrual migraine by ICHD criteria

Exclusion Criteria:

1. Not actively practicing adequate contraception or intending to continue to do so during the treatment.
2. 15 or more days of headache during each of the prior 3 months
3. Prior use of Treximet for the treatment of menstrual migraine
4. Uncontrolled hypertension
5. Hemiplegic or basilar migraine
6. Clinical evidence of coronary artery disease or other clinically significant and relevant cardiac disease (e.g. vasospastic angina)
7. History of stroke or transient ischemic attack
8. History of ischemic bowel disease
9. Clinically significant hepatic disease
10. History of allergy to any NSAID or triptan
11. History of gastritis, peptic ulcer disease, GI bleeding, gastric surgery

Min Age: 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2011-01; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Total dose of study medication | 90 days
  Endpoints will include (a) total doses of study medication taken (primary endpoint), (b) total doses of rescue medication taken, (c) total "migraine days", (d) total "headache days", (e) days of functionally incapacitating headache, (f) work-related absenteeism, (g) unscheduled visits for acute headache treatment, (h) cost of unscheduled visits for acute headache treatment, (i) safety and tolerability, and (j) patient satisfaction.

SECONDARY OUTCOMES:
total doses of rescue medication taken | 90 days
  The participant records in the diary how many doses of the rescue medication has been taken since their last visit
total "headache days" | 90 days
  The participant records in their diary how many headache days the participant has had since their last visit.
days of functionally incapacitating headache | 90 days
  The participant records in the diary how many of their headache days consisted of functionally incapacitating headaches.
work-related absenteeism | 90 days
  The particpant records in their diary how many of the headaches caused work-related absences.
unscheduled visits for acute headache treatment | 90 days
  The participant records in their diary how many unscheduled visits have occurred due to acute headache treatment
cost of unscheduled visits for acute headache treatment | 90 days
  The participant records in their diary how many unscheduled visits and the cost of each that occurred due to acute headache treatments.
safety and tolerability | 90 days
  determine the saftety and the tolerability of the study medication at time of visit or as reported prior to visit via participant report of side effects or adverse events.
patient satisfaction | 90 days
  determine participant's satisfaction with her ability to manage the cycle of MM as measured by a 5 point Likert scale.

CONTACTS AND LOCATIONS:
Overall Officials: J Ivan Lopez, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States